CLINICAL TRIAL: NCT05482347
Title: Development of a Decision Aid for Parents of Children With Neurogenic Bladder Considering Surgical Reconstruction
Brief Title: Educational Video for Neurogenic Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-1926
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Neurogenic Bladder
MeSH Terms: conditions — Urinary Bladder, Neurogenic

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants will be masked to which arm of the study to which they are randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (knowledge assessment before video) (Active Comparator): The patient will complete the knowledge assessment, then they will be presented with the educational video. After watching the video, they will complete the acceptability scale questionnaire and will be asked to select a gift card preference at the end of the survey.
  Interventions: Other: Educational video
- Video (video before knowledge assessment) (Experimental): The patient will be presented with the educational video, then they will complete the knowledge assessment and the acceptability scale questionnaire. They will be asked to select a gift card preference at the end of the survey.
  Interventions: Other: Educational video

INTERVENTIONS:
Other: Educational video — The intervention is an educational video developed using data from focus groups of families with children diagnosed with neurogenic bladder.

SUMMARY:
This study is designed to assess the efficacy of educational materials in parents of children with neurogenic bladder considering surgical reconstruction. Focus groups were conducted with neurogenic bladder patients and their families in which participants were asked questions about expectations, fears, medical understanding, unexpected challenges, and persistent questions regarding reconstructive surgery for neurogenic bladder. Analysis of this qualitative data was used to create educational materials (such as animated videos) and decision-making tools for families of children with neurogenic bladders who are trying to decide what treatment option is right for them, and to better prepare them for what lies ahead. This study specifically aims to investigate the effect of an educational video on participants' knowledge of neurogenic bladder and surgical management.

DETAILED DESCRIPTION:
Within pediatric urology, some of the most complex and consequential decision-making surrounds surgical management of the neurogenic bladder. There is strong evidence that more informed patients are more adherent, more engaged, more likely to fully consider the risks and benefits of different treatment options, and ultimately more satisfied with their clinical outcome. In practice, patient education is time-consuming, inconsistent, and often complicated by language barriers and varying levels of medical literacy. A potential solution to overcoming the barriers to educating patients and families on these complex issues lies in patient decision aids and quality medical educational videos.

The investigators, using qualitative data obtained from focus groups with patient families, developed an educational video on neurogenic bladder for patients and their families. This study will assess the efficacy of the educational video by utilizing a knowledge questionnaire that is administered to participants who have been and who have not been exposed to the video. The investigators will identify all patients between the ages of 0 and 18 years old who have a diagnosis of neurogenic bladder, but have not undergone any surgical treatment for neurogenic bladder. All eligible patients' caregivers will be invited to participate in this study, which will be administered virtually via a REDCap survey that is disseminated by email. Patients' caregivers will provide consent electronically, after which they will be randomized into a control or intervention arm. Randomization will be stratified by age groups (0-4 years, 5-11 years, and 12 years and older). These age groups were defined based on patients' independence regarding ability to manage their diagnosis (i.e., 0-4 years represents patients before toilet training; 5-11 years represents patients who are school-aged but still require adult supervision; and 12 years and older represents patients who have relatively increased independence). Participants in the control arm will take the knowledge questionnaire, then watch the educational video, while participants in the intervention arm will watch the educational video prior to taking the knowledge questionnaire. Both groups will be asked to provide feedback on the educational video afterwards. The investigator will determine the average knowledge questionnaire score within each group (control and intervention) and compare the two averages.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking parents/and or primary caregivers of children 18 years old or younger with a diagnosis of neurogenic bladder who have received care at Children's Hospital Colorado, but have not undergone a major surgery for the treatment of neurogenic bladder

Exclusion Criteria:

* Parent/caregiver does not speak English
* Children who have undergone a major surgery for the treatment of neurogenic bladder (ex. urinary diversion)
* Patients greater than 18 years old

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Comparison of average knowledge assessment scores between participants in the intervention group compared participants to the control group | End of study (6 months)
  The knowledge assessment consists of 6 multiple choice questions, each with 4 answer choices, regarding participants' knowledge on the condition of neurogenic bladder. The questionnaire will be scored based on how many questions the participants correctly answer and an average score will be calculated for the intervention group and the control group. Average scores for each of the predefined age groups will also be calculated and compared within the control and intervention groups.

SECONDARY OUTCOMES:
Acceptability of educational video | End of study (6 months)
  The acceptability scale consists of 12 questions (multiple choice questions, free responses, and rating questions) asking participants for feedback regarding the educational video, as well as suggestions on how to improve the video for future patients. One question, formatted as a yes/no question, will be used to assess the acceptability of the education video and asks participants if they would recommend the educational video to other parents/families of children with neurogenic bladder at different times over the course of diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Buchanan, PhD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No